CLINICAL TRIAL: NCT00059228
Title: The Efficacy of 17Beta-Estradiol in Postpartum-Related Depressive Illness
Brief Title: Clinical Trial of Estrogen for Postpartum Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 030161; 03-M-0161
Record Dates: First submitted 2003-04-22; First posted 2003-04-22 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Postpartum Depression; Depression
Keywords: Pregnancy; Gonadal Steroids; Antidepressants; Puerperium; Depression; Postpartum; Estradiol; Estrogen Response Element; Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum; Depression | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Estradiol (Experimental): Experimental
  Interventions: Drug: 17beta Estradiol
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: 17beta Estradiol — Alora 100 microgram per day by skin patch for 6 weeks.
  Arms: Estradiol
Drug: Placebos — Placebo skin patch for 6 weeks
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of estrogen treatment in women with postpartum depression (PPD).

PPD causes significant distress to a large number of women; the demand for effective therapies to treat PPD is considerable. Estradiol therapy has a prophylactic effect in women at high risk for developing PPD. The prevention of a decline in estradiol levels may prevent the onset of PPD. Studies also suggest that estradiol has antidepressant effects in women and may provide a safe and effective alternative to traditional antidepressants in women with PPD.

Participants will be screened with a medical history, physical examination, blood and urine tests, psychological tests, genetic studies, and self-rating scales and questionnaires. Upon study entry, women will be randomly assigned to wear skin patches containing either estradiol or placebo (a patch with no active ingredient) for 6 weeks. Women who receive estradiol and do not menstruate during the last week of the study will receive progesterone for 7 days to initiate menstruation. Women who receive placebo and do not menstruate during the last week of the study will continue to receive placebo at the end of the study. Every week, participants will have blood taken and will be asked to complete symptom self-rating scales. A urine sample and blood samples will be collected at different time points through out of the study. Participants who receive placebo and those whose symptoms do not improve with estradiol therapy will be offered treatment with standard antidepressant medications for 8 weeks at the end of the study.

DETAILED DESCRIPTION:
Postpartum-related mood disorders cause significant distress to a potentially large number of women. The demand for effective therapies for treating these mood disorders is considerable, as is the need to define clinical or biologic markers that may predict successful response of these mood disturbances to estradiol. Despite the prevalence of postpartum depressions, only a few double-blind, controlled trials of antidepressant agents have been performed in this condition (1-4)- only two of which were placebo-controlled. A recent large multicenter trial failed to confirm the initially promising but anecdotal reports of the protective role of fish oil in PPD (5). Similarly, despite evidence of estradiol s therapeutic efficacy in trials

that were both open (monotherapy) (6) and controlled (combined with traditional antidepressant agents (7)), the potential of estradiol to be an effective alternative to traditional psychotropics in postpartum depression has not been examined under controlled conditions.

Postpartum depressions occur by definition after delivery when women are relatively hypogonadal. Indeed, plasma estradiol and progesterone levels are low and comparable to those seen during the peri and postmenopause. However, there is no evidence that postpartum depression represents a simple hormone deficiency, and women with postpartum depression are not distinguished from women without postpartum depression on the basis of any abnormality of basal reproductive hormones. Nonetheless, a role for declining estradiol secretion has been suggested by the following observations: 1) estradiol therapy has been reported to have a prophylactic effect in women at high risk for developing postpartum depression (8), suggesting that the prevention of a decline in estradiol levels (threshold or rate of decline) may prevent the onset of postpartum depression in some women; and (2) declining ovarian steroids trigger the onset of mood disturbances in women with but not women without a history of postpartum depression during a scaled down model of pregnancy in the puerperium (9). Thus, as with depressions occurring during the perimenopause, when ovarian hormone secretion is also declining, postpartum depression may also be responsive to estradiol therapy. In fact, open trials of estradiol therapy in postpartum depression (6) as well as a trial of estradiol in combination with traditional antidepressants (7) have suggested that estradiol does have antidepressant-like effects that are observed within a three week time period in women with postpartum onset major depression. Thus, estradiol treatment may not only provide a safe and effective alternative to traditional antidepressants in women with postpartum depression, but it may also suggest the relevant hormonal trigger for the development of this condition.

In this protocol we wish to investigate the effects of estradiol on mood in women with moderately severe postpartum depression under placebo controlled conditions. This protocol will address the following question: 1) Does estradiol improve mood in postpartum depressed women?

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. A history of at least two weeks with postpartum-related mood disturbances of moderate severity, and self-report of the onset of depression within three months of a normal vaginal delivery or uncomplicated Caesarean section;
  2. A current episode of minor (meeting 3-4 criterion symptoms) or major depression (of moderate severity or less on the SCID severity scale and not meeting DSM-IV criteria symptom 9 [suicidal ideation]) as determined by the administration of the minor depression module of the SADS-L and the Structured Clinical Interview for DSM-IV. Additionally, to ensure that subjects meet a minimum threshold for severity of depression, subjects will have scores greater than or equal to 10 on either the Beck Depression Inventory (BDI) or the Center for Epidemiologic Studies - Depression (CES-D) Scale during at least three of the six clinic visits during the two week screening phase, as well as a 17 item Hamilton Depression score greater than or equal to 10. Subjects will be excluded if they meet any of the following criteria: major depression of greater than moderate severity (including postpartum psychosis). DSM-IV criteria #9 (suicidal ideation), or anyone requiring immediate treatment after clinical assessment.
  3. Not greater than six months post delivery;
  4. Age 20 to 45;
  5. In good medical health, and not taking any medication or dietary and herbal supplements on a regular basis (with the exception of multivitamins or calcium supplements).

EXCLUSION CRITERIA:

The following conditions will constitute contraindications to treatment and will preclude a subject s participation in this protocol:

1. severe major depression with any of the following:

   * positive (threshold) response to SCID major depression section item # 9, suicidal ideation;
   * anyone requiring immediate treatment after clinical assessment;
   * severity ratings greater than moderate on the SCID IV interview (including postpartum psychosis);
2. current treatment with antidepressant medications
3. history of psychiatric illness during the two years before the reported onset of the current episode of depression or a history of either mania (DSM-IV criteria) or postpartum psychosis at any time in the past.
4. history of ischemic cardiac disease, pulmonary embolism, retinal thrombosis, or thrombophlebitis; any subject with risk factors for thrombo-embolic phenomena including cigarette smokers (greater than 10 cigarettes per day), varicose veins, patients with prolonged periods of immobilization (including prolonged travel), and active heart disease.
5. renal disease, asthma
6. hepatic dysfunction
7. women with a history of carcinoma of the breast, or women with a family history of the following: premenopausal breast cancer or bilateral breast cancer in a first degree relative; multiple family members (greater than three relatives) with postmenopausal breast cancer
8. women with a history of uterine cancer, endometriosis, ill-defined pelvic lesions, particularly undiagnosed ovarian enlargement, undiagnosed vaginal bleeding
9. patients with a known hypersensitivity to estradiol, transdermal skin patches, or medroxyprogesterone acetate
10. pregnant women
11. porphyria
12. diabetes mellitus
13. cholecystitis or pancreatitis
14. history of cerebrovascular disease (stroke), epilepsy, hypertension, hypercalcemia
15. recurrent migraine headaches
16. malignant melanoma
17. history of familial hyperlipoproteinemia
18. prior hormonal therapy for the treatment of postpartum-related mood or physical symptoms within the last six months
19. history of psychiatric illness during the two years prior to the reported onset of the current episode of depression

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2003-04-17; Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ahokas A, Kaukoranta J, Wahlbeck K, Aito M. Estrogen deficiency in severe postpartum depression: successful treatment with sublingual physiologic 17beta-estradiol: a preliminary study. J Clin Psychiatry. 2001 May;62(5):332-6. doi: 10.4088/jcp.v62n0504. PMID 11411813
- [Background] Gregoire AJ, Kumar R, Everitt B, Henderson AF, Studd JW. Transdermal oestrogen for treatment of severe postnatal depression. Lancet. 1996 Apr 6;347(9006):930-3. doi: 10.1016/s0140-6736(96)91414-2. PMID 8598756
- [Background] Bloch M, Schmidt PJ, Danaceau M, Murphy J, Nieman L, Rubinow DR. Effects of gonadal steroids in women with a history of postpartum depression. Am J Psychiatry. 2000 Jun;157(6):924-30. doi: 10.1176/appi.ajp.157.6.924. PMID 10831472

RESULTS

PARTICIPANT FLOW:
Groups:
- Estradiol: Estradiol transdermal patch 100mcg
- Placebo: Placebo transdermal patch
Period: Overall Study
Arm/Group | Estradiol | Placebo
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory
Description: The Beck Depression Inventory (BDI) is a 21-question multiple-choice self-report inventory for measuring the severity of depression. Higher total scores indicate more severe depressive symptoms. The range of scores vary from 0 to 63 (highest possible total) for the whole test. A score of 0 - 10 indicates minimal depression, while a score of over 40 indicates extreme depression. No subscales were used for this outcome.
Time Frame: 6 weeks
Population: The analysis included only those subjects who had taken Estradiol and Placebo
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 6 | 6
Units on a scale | 15.84 (3.91) | 5.3 (3.19)

2. Primary Outcome: Beck Depression Inventory
Description: as for outcome 1
Time Frame: Baseline
Population: The analysis included only those subjects who had taken Estradiol and Placebo
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | 26 (2.62) | 27.67 (3.72)

ADVERSE EVENTS:
Arm/Group | Estradiol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol (N=6) | Placebo (N=6)
Nausea (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes